CLINICAL TRIAL: NCT04320732
Title: Risk Factors for Community- and Workplace Transmission of COVID-19
Status: Recruiting | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: Age Labs AS (Unknown)
Responsible Party: Principal Investigator, Arne Vasli Lund Søraas, Principal Investigator, MD, PhD, Oslo University Hospital
Other Study IDs: REK-124170
Record Dates: First submitted 2020-03-23; First posted 2020-03-25 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-11

CONDITIONS: Coronavirus
MeSH Terms: conditions — Coronavirus Infections | interventions — Behavior Observation Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and upper repiratory samples will be collected from some participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Individuals with COVID-19 infection: Confirmed by routine laboratory diagnosis. All types of COVID-19 disease from asymptomatic carriers to hospitalized patients can be included.
  Only subjects >18 years old will be included in the study.
  Interventions: Behavioral: Observation of behavior and COVID-19 infection will be conducted.
- Individuals tested for COVID-19 infection with negative test: Confirmed by routine laboratory diagnosis
  Interventions: Behavioral: Observation of behavior and COVID-19 infection will be conducted.
- Healthy individuals: Recruitet from the general population
  Interventions: Behavioral: Observation of behavior and COVID-19 infection will be conducted.
- Risk groups for COVID-19 exposure: Including, but not limited to healthcare workers.
  Interventions: Behavioral: Observation of behavior and COVID-19 infection will be conducted.
- Patients admitted to hospital: Without COVID-19 infection.
  Interventions: Behavioral: Observation of behavior and COVID-19 infection will be conducted.

INTERVENTIONS:
Behavioral: Observation of behavior and COVID-19 infection will be conducted. — No intervention, only prospective observation of behavior will be conducted by a questionnaire.

SUMMARY:
The project is an epidemiological observational study based on an electronic questionnaire on risk factors for COVID-19 in the community and healthcare setting.

DETAILED DESCRIPTION:
Summary The data collected will identify real-life risk factors for getting the COVID-19 diagnosis.

The Oslo University Hospital/University of Oslo web-based solution "nettskjema" will be used to collect data and consent forms.

The impact of knowing the risk factors for COVID-19 is tremendous because it can enable governments to conduct more targeted public health measurements than today to reduce the spread of the virus.

Detailed description Research into an ongoing COVID-19 outbreak is difficult because patients are isolated, and supplies of personal protective equipment (PPE) supplies are limited. The risk of transmission to study personal is non-negligible even when PPE is available.

A study design based on an electronic questionnaire and consent from delivered from the Oslo University Hospital/University of Oslo, GDPR (General Data Protection Regulation) compliant "TSD" service has therefore been chosen.

The study will be a case-control study based on a combined electronic consent form and questionnaire that the participants will fill in using a smartphone and electronic identification.

The groups that will be included are:

* Hospitalized and non-hospitalized patients/persons with COVID-19 at all stages of the disease and after the disease
* Hospitalized patients without COVID-19
* Healthcare personal or other groups with an increased risk of COVID-19
* Healthy volunteers

Participants may be followed with repeated questionnaires prospectively.

Biological samples Biological samples may hold crucial information about the susceptibility to COVID-19 and for susceptibility to the progression of the disease. It is within the scope of the study to analyze such samples from a limited number of participants which will be asked to provide such samples or hospitalized patients that have surplus material. The material will be analyzed with non-genetic methods most suitable to provide such information.

ELIGIBILITY:
Inclusion Criteria:

* Norwegian adult

Exclusion Criteria:

* Unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will be a combined retrospective and prospective case-control study based on a combined electronic consent form and questionnaire that the study groups will fill in using a smartphone and electronic identification.
  The groups that will be included are:
  * Hospitalized and non-hospitalized patients/persons with COVID-19 at all stages of the disease and after the disease
  * Hospitalized patients without COVID-19
  * Healthcare personal or other groups with an increased risk of COVID-19
  * Healthy volunteers
  Probability sampling will be conducted, but not solely.
Sampling Method: Probability Sample
Enrollment: 250000 (Estimated)
Dates: Start 2020-03-27 (Actual); Primary Completion 2025-03-27 (Estimated); Study Completion 2030-03-20 (Estimated)

PRIMARY OUTCOMES:
Rate of COVID-19 infection | 1 year
  Diagnosed with serology or direct viral detection

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
European GDPR regulations severely limits IPD, but the study will share data to the largest extent possible within GDPR.